CLINICAL TRIAL: NCT04714047
Title: Progressive Resistance Training Compared to Neuromuscular Exercise in Patients With Hip Osteoarthritis, and the Additive Effect of Booster Sessions: A Multicenter Randomized Controlled Trial
Brief Title: Progressive Resistance Training Compared to Neuromuscular Exercise in Patients With Hip Osteoarthritis
Acronym: HipBooster
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Vejle Hospital (Other); Naestved Hospital (Other); Regional Hospital Holstebro (Other); Aarhus University Hospital (Other); Physiotherapy Associates (Other); Slagelse Hospital (Other); University of Southern Denmark (Other); Regionshospitalet Silkeborg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HipBooster
Record Dates: First submitted 2021-01-15; First posted 2021-01-19 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2023-05

CONDITIONS: Hip Osteoarthritis
Keywords: Progressive Resistance Training; Neuromuscular Exercise; Physical Therapy; Physical Rehabilitation
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: (Experimental): PRT
  Interventions: Other: Progressive Resistance Training and no booster sessions
- Group 2: (Experimental): PRT + Booster sessions
  Interventions: Other: Progressive Resistance Training and booster sessions
- Group 3: (Active Comparator): NEMEX
  Interventions: Other: Neuromuscular exercise and no booster sessions
- Group 4: (Experimental): NEMEX + Booster sessions
  Interventions: Other: Neuromuscular exercise and booster sessions

INTERVENTIONS:
Other: Progressive Resistance Training and no booster sessions — An initial 12-week exercise intervention, consisting of 1-hour group sessions of progressive resistance training supervised by a physiotherapist 2 times per week.
  The sessions consist of a 10-minute submaximal warm up on an exercise bike followed by 50 minutes of PRT with exercises targeting the muscles of the hip and knee joints; leg press, hip extension, hip abduction, hip flexion and knee extension. The progression will be in line with guidelines provided by the American College of Sports Medicine. The intensity will follow repetition maximum (RM) targets, from 12 RM for the first week towards 8 RM for the last weeks.
  After the 12 weeks, this group consists of patients who are randomized to receive no further treatment. For the following 9 months, these patients are given a membership to a fitness center where they are encouraged to continue the same exercise regime.
  Arms: Group 1:
Other: Progressive Resistance Training and booster sessions — An initial 12-week exercise intervention, consisting of 1-hour group sessions of progressive resistance training supervised by a physiotherapist 2 times per week.
  The sessions consist of a 10-minute submaximal warm up on an exercise bike followed by 50 minutes of PRT with exercises targeting the muscles of the hip and knee joints; leg press, hip extension, hip abduction, hip flexion and knee extension. The progression will be in line with guidelines provided by the American College of Sports Medicine. The intensity will follow repetition maximum (RM) targets, from 12 RM for the first week towards 8 RM for the last weeks.
  After the 12 weeks, this group consists of patients who are randomized to receive 4 booster sessions (at 1, 3, 5 and 7 months after termination of the initial 12 week intervention). Additionally, for the following 9 months, these patients are given a membership to a fitness center where they are encouraged to continue the same exercise regime without supervision.
  Arms: Group 2:
Other: Neuromuscular exercise and no booster sessions — An initial 12-week exercise intervention, consisting of 1-hour group sessions of progressive resistance training supervised by a physiotherapist 2 times per week.
  The sessions consist of a 10-minute submaximal warm up on an exercise bike followed by 50 minutes of NEMEX training with exercises focused on stability, postural function, postural orientation, lower extremity muscle strength, and functional exercises. Progression is made when an exercise is performed with good sensorimotor control and good quality of the performance and with minimal exertion and adequate control of the movement.
  After the 12 weeks, this group consists of patients who are randomized to receive no further treatment. For the following 9 months, these patients are given equipment and encouraged to continue the same exercise regime at home without supervision.
  Arms: Group 3:
Other: Neuromuscular exercise and booster sessions — An initial 12-week exercise intervention, consisting of 1-hour group sessions of progressive resistance training supervised by a physiotherapist 2 times per week.
  The sessions consist of a 10-minute submaximal warm up on an exercise bike followed by 50 minutes of NEMEX training with exercises focused on stability, postural function, postural orientation, lower extremity muscle strength, and functional exercises. Progression is made when an exercise is performed with good sensorimotor control and good quality of the performance and with minimal exertion and adequate control of the movement.
  After the 12 weeks, this group consists of patients who are randomized to receive 4 booster sessions (at 1, 3, 5 and 7 months after termination of the initial 12 week intervention). Additionally, for the following 9 months, these patients are given equipment and encouraged to continue the same exercise regime at home.
  Arms: Group 4:

SUMMARY:
The primary aim of this randomized controlled trial is to investigate the effectiveness of 12 weeks of progressive resistance training (PRT) compared to neuromuscular exercise (NEMEX) on functional performance in patients with hip OA measured by the 30-seconds chair stand test. Secondary aims are to investigate; the determinants of improvement in physical function following PRT or NEMEX; the effectiveness of booster sessions in prolonging the effects of the initial interventions (12 months), the cost-effectiveness of booster sessions (12 months). We will test the hypothesis that PRT is superior to NEMEX in improving physical function measured with the 30s sit-to-stand test at 12 week follow-up.

DETAILED DESCRIPTION:
This randomized controlled trial will be a multicenter trial involving hospitals and physiotherapy clinics across Denmark. Part 1: For the initial 12-week exercise intervention, participants will be randomized into two groups: PRT or NEMEX. Part 2: After the initial intervention, participants in each group will be randomized to booster sessions (PRT+B and NEMEX+B) or to receive no further treatment (PRT-B and NEMEX-B). Booster sessions will be provided at 4, 6, 8 and 10 months after baseline. Outcomes will be measured at baseline, after 12 weeks of intervention, and at 6-, 9- and 12-months follow-up.

The exercise interventions will be performed at the collaborating hospitals and physiotherapy clinics across Denmark. All sessions will be conducted in group sessions with one physiotherapist supervising the exercises. The duration and frequency of the interventions will be 12 weeks with 2 supervised sessions each week. If participants experience pain during exercise exceeding 5 out of 10 on a Visual Analogue Scale (VAS), the physiotherapist will modify the exercise, decreasing the exercise intensity (load) or modifying the range of motion. All unilateral exercises will be performed for both sides.

The NEMEX intervention will follow the NEMEX program as described by Ageberg et al. The sessions consist of a 10-minute submaximal warm up on an exercise bike followed by 50 minutes of NEMEX training with exercises focused on stability, postural function, postural orientation, lower extremity muscle strength, and functional exercises.

The PRT intervention will follow the same protocol for training frequency and duration as the NEMEX intervention. The sessions consist of a 10-minute submaximal warm up on an exercise bike followed by 50 minutes of PRT with exercises targeting the muscles of the hip and knee joints; leg press, hip extension, hip abduction, hip flexion and knee extension.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed OA of the hip joint according to the National Institute for Health and Care Excellence criteria
* Have experienced pain of at least 3 out of 10 on the visual analog scale in the index hip within the last two weeks
* Age ≥ 45 years
* No surgery in the lower extremities six months prior to inclusion
* No comorbidity that prevents exercising
* Adequacy in written and spoken Danish
* Not being a candidate for total hip arthroplasty

Exclusion Criteria:

* BMI score > 40
* Pregnancy
* Resistance training or neuromuscular training for the lower extremities for more than 12 sessions in the last 6 months or 6 sessions in the last 3 months (resistance training is defined by the American College of Sports Medicine guidelines while neuromuscular training is defined by exercises involving multiple joints and muscle groups performed in functional weight-bearing positions with emphasis on the quality and efficiency of movement, as well as alignment of the trunk and lower limb joints)
* Planned vacation for more than 14 days within the 12-week intervention period without the possibility of expanding the intervention accordingly

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-03 (Actual)

PRIMARY OUTCOMES:
Change in functional performance measured by the 30-seconds chair stand test | Measured at baseline, 12 week and 12 month follow-up.
  The 30-second chair stand test is a valid and responsive measure of lower-extremity muscle strength evaluating sit-to-stand function, which is limited in people with lower extremity OA.

SECONDARY OUTCOMES:
Change in 40m fast-paced walk test | Measured at baseline, 12 week and 12 month follow-up.
  Time (in seconds) taken to complete a 40 m course at fast walking pace.
Change in 9 step stair climb test | Measured at baseline, 12 week and 12 month follow-up.
  Time (in seconds) taken to negotiate 9 steps on a standard step-height stair-way (up and down).
Change in leg extension muscle power (watt/kg bodyweight) | Measured at baseline, 12 week and 12 month follow-up.
  Leg extensor muscle power (force times acceleration) will be measured using the Nottingham Power Rig (NPR). The NPR measures the power output in total watt and watt pr. bodyweight in kilograms from a seated push on a flat pedal which is transmitted by a lever and chain to spin a flywheel. The NPR is a safe and reliable method to measure explosive knee extensor muscle power and has been validated as a clinically important measure of muscle function in elderly individuals.
Change in the HOOS pain subscale | Measured at baseline, 12 week and 12 month follow-up.
  The HOOS pain subscale is a 10-item patient-reported outcome measure designed to assess other hip symptoms in patients with hip osteoarthritis. The total score ranges from 0 to 100, with higher scores indicating better symptoms status.
Change in the HOOS activities of daily living (ADL) function subscale | Measured at baseline, 12 week and 12 month follow-up.
  The HOOS ADL function subscale is a 17-item patient-reported outcome measure designed to assess ADL function in patients with hip osteoarthritis. The total score ranges from 0 to 100, with higher scores indicating better ADL function status.
Change in the HOOS quality-of-life subscale | Measured at baseline, 12 week and 12 month follow-up.
  The HOOS quality-of-life subscale is a four-item patient-reported outcome measure designed to assess hip-related quality-of-life in patients with hip osteoarthritis. The total score ranges from 0 to 100, with higher scores indicating better quality-of-life status.
Change in the HOOS sports and recreation subscale | Measured at baseline, 12 week and 12 month follow-up.
  The HOOS sports and recreation subscale is a four-item patient-reported outcome measure designed to assess sports and recreation function in patients with hip osteoarthritis. The total score ranges from 0 to 100, with higher scores indicating better sports and recreation status.
Global Perceived Effect (GPE) | Measured at 12 week and 12 month follow-up.
  The GPE of the interventions will be assessed for three domains on a 7-point Likert scale
Change in muscle strength | Measured at baseline, 12 week and 12 month follow-up.
  Muscle strength is measured in a standardized one-repetition maximum test for the leg press exercise.
Change in the HOOS symptoms subscale | Measured at baseline, 12 week and 12 month follow-up.
  The HOOS symptoms subscale is a five-item patient-reported outcome measure designed to assess hip symptoms in patients with hip osteoarthritis. The total score ranges from 0 to 100, with higher scores indicating better symptoms status.
Adherence to the 12 week initial intervention | Registered throughout the 12 week initial intervention.
  High adherence is defined as ≥ 80% attendance to the supervised interventions.
Adherence to the 9 months of self-administered training | Registered throughout the 9 months follow-up period.
  High adherence is defined by ≥ 80% of the assigned exercise programs performed at home or at the fitness center.
AE (Adverse Events) & Serious Adverse Events (SAE) | Registered throughout the 12 month study period.
  Continous registration of health issues and injuries. Physiotherapists in charge of the training sessions will monitor potential AE and SAE. Also, during the follow-up visits at week 12 and 12 months, the participants will be asked about potential AE's and SAE's using open-probe questions.
Drop-outs | Registered throughout the 12 month study period.
  Number og drop-out from the training interventions.

OTHER OUTCOMES:
Number of joint replacements | Measured at baseline and 12 month follow-up.
  Patient-reported joint replacements
Productivity Costs Questionnaire (IPCQ) | Measured at 12 week and 6, 9, 12 month follow-up.
  The IPCQ questionnaire includes three modules measuring productivity losses of paid work due to 1) absenteeism and 2) presenteeism and productivity losses related to 3) unpaid work
Physical activity level | Measured at baseline, 12 week and 12 month follow-up.
  Patient reported physical activity levels is assessed with a three domain questionnaire.
Change in pain measured on a Numerical Rating Scale (NRS) | Measured at baseline, 12 week and 12 month follow-up.
  NRS pain score will be measured before and after each exercise session and at each follow-up evaluation before and after completing the functional performance tests.
Healthcare Utilization Questionnaire (HUQ) | Measured at baseline, 12 week and 6, 9, 12 month follow-up.
  The HUQ is a nine-item patient-reported outcome measure designed to assess healthcare and medicine usage.
Change in EuroQol Group 5-dimension 5-level (EQ-5D-5L) | Measured at baseline, 12 week and 6, 9, 12 month follow-up.
  The EQ-5D-5L is a five-item patient-reported outcome measure designed to assess generic health-related quality-of-life. The total score of the descriptive index and EQ-VAS ranges from -0.624 (worst) to 1.000 (best) and 0 (worst imaginable health) to 100 (best imaginable health), respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Troels Kjeldsen, MSd, Principal Investigator — Aarhus University Hospital and Aarhus University; Inger Mechlenburg, Prof., Study Director — Aarhus University Hospital and Aarhus University; Søren T Skou, Prof., Study Director — Slagelse Hospital and University of Southern Denmark; Ulrik Dalgas, Prof., Study Director — University of Aarhus
Locations (3):
- Denmark (3):
  - Aarhus University, Aarhus
  - Aarhus University Hospital, Aarhus N
  - Næstved-Slagelse-Ringsted Hospitals, Slagelse

IPD SHARING:
Plan to Share IPD: Yes
Anonymised patient-level data for the primary and all secondary outcome measures will be made available if required by the scientific journal, in which the results of the trial are published.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available after publication of the trial.
Access Criteria: Data access will be reviewed by the author group. Requesters will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Kjeldsen T, Dalgas U, Skou ST, Tonning LU, Ingwersen KG, Birch S, Holm PM, Garval M, Varnum C, Callesen J, Foldager F, Bibby BM, Mechlenburg I. Booster sessions for maintaining the effect of neuromuscular exercise and progressive resistance training in hip osteoarthritis: 12-month follow-up from a multicenter cluster-randomized controlled trial. Osteoarthritis Cartilage. 2025 Nov;33(11):1393-1403. doi: 10.1016/j.joca.2025.07.012. Epub 2025 Jul 23. PMID 40712915
- [Derived] Kjeldsen T, Skou ST, Dalgas U, Tonning LU, Ingwersen KG, Birch S, Holm PM, Frydendal T, Garval M, Varnum C, Bibby BM, Mechlenburg I. Progressive Resistance Training or Neuromuscular Exercise for Hip Osteoarthritis : A Multicenter Cluster Randomized Controlled Trial. Ann Intern Med. 2024 May;177(5):573-582. doi: 10.7326/M23-3225. Epub 2024 Apr 9. PMID 38588540
- [Derived] Kjeldsen T, Dalgas U, Skou ST, van Tulder M, Bibby BM, Mechlenburg I. Progressive resistance training compared to neuromuscular exercise in patients with hip osteoarthritis and the additive effect of exercise booster sessions: protocol for a multicentre cluster randomised controlled trial (The Hip Booster Trial). BMJ Open. 2022 Sep 15;12(9):e061053. doi: 10.1136/bmjopen-2022-061053. PMID 36109033

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT04714047/SAP_000.pdf